CLINICAL TRIAL: NCT07361562
Title: A Study of a Selective ERBB2 Inhibitor, CGT4255, in Patients With Advanced Solid Tumors With ERBB2 Genetic Alterations or HER2 Overexpression
Brief Title: A Study of a Selective ERBB2 Inhibitor (CGT4255), in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CGT4255-25-101
Record Dates: First submitted 2025-12-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor, Adult; ERBB2 Altered Breast Cancer; ERBB2 Gene Amplification; HER2 Overexpression; Non-Small Cell Lung Cancer; HER2
Keywords: ERBB2 genetic alterations; Investigational Drug; Advanced Solid Tumors; ERBB2 Mutated Non Small Cell Lung Cancer; Mutated Advanced Solid Tumors; ERBB2 Brain Metastases; ERRB2 Point Mutations; ERBB2 Gene Short Variants; ERBB2 Gene Rearrangements; ERBB2 activation alteration; ERBB2 gene copy number amplifications; ERBB2 gene insertions; ERRB2 gene deletions; ERBB2 gene fusions; NRG1 gene fusions; ERBB2 indel; Phase 1/1b; HER2 Protein Overexpression; HER2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Phase 1, Part A evaluating multiple ascending doses.
  Phase 1b, evaluation of Part A selected doses in 2 cohorts defined by tumor type including a randomized dose optimization design (Part B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Part A: Dose Escalation Multiple doses of CGT4255 for oral administration
  Interventions: Drug: CGT4255
- Signal Seeking and Dose Escalation (Experimental): Part B: Signal Seeking and Dose Optimization Oral dose(s) of CGT4255 at the selected dose levels determined in Phase 1
  Interventions: Drug: CGT4255
- Signal Seeking (Experimental): Part C: Includes signal seeking. Participants will receive CGT4255 at a dose level selected based on data from Part A
  Interventions: Drug: CGT4255

INTERVENTIONS:
Drug: CGT4255 — CGT4255 Daily Oral Administration

SUMMARY:
This is an open-label, phase 1/1b study evaluating the safety, tolerability, pharmacokinetic (what the body does to the drug), pharmacodynamic (what the drug does to the body), and antitumor activity of CGT4255 in adult participants with advanced solid tumors with ERBB2 alterations or HER2 overexpression.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed diagnosis of:

   1. Part A: Locally advanced, metastatic, and/or unresectable solid tumor with documented ERBB2-activating alteration or NRG1 gene fusion in blood and/or tumor or HER2 overexpression in tumor
   2. Part B: Locally advanced, metastatic, and/or unresectable NSCLC with documented ERBB2 mutation in blood and/or tumor
   3. Part C: Locally advanced, metastatic and/or unresectable breast cancer with documented ERBB2 mutation in blood and/or tumor or HER overexpression in tumor
2. Have measurable disease per RECIST v1.1.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1 for Part A. For Parts B and C, ECOG Performance Status must be 0 to 2.
4. Have clinically acceptable local laboratory screening results (clinical chemistry and hematology) within certain limits.

Exclusion Criteria:

1. Received small molecule chemotherapy or anticancer therapies or radiotherapy within certain timeframes before first dose of study drug.
2. Major surgeries (eg, craniotomy and thoracotomy) within 4 weeks of the first dose of study drug.
3. Treatment with palliative focal radiotherapy (cranial or extracranial) (eg, stereotactic radiosurgery or intensity-modulated radiation therapy) ≤2 weeks before the first dose of study drug; treatment with whole-brain radiotherapy ≤4 weeks before the first dose of study drug.
4. Clinically significant cardiac disease.
5. Resolution of toxicities from prior therapy to ≤Grade 1 (or baseline), including resolution of clinically significant laboratory abnormalities, before the first dose of study drug.
6. Restrictions on use of corticosteroid use to manage neurologic symptoms in different parts of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) [Part A] | Approximately 12 months
  1. Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) and AEs leading to dose modifications and dose limiting toxicities (DLTs) to determine the maximum tolerated dose (MTD) or the maximum evaluated dose (MED) in participants with ERBB2-altered advanced solid tumors
Overall Response Rate [Part B and Part C] | Approximately 6 months
  Overall Response Rate (ORR), determined by confirmed CR + PR of all lesions (intracranial and extracranial), based on Investigator assessment using the whole-body RECIST v1.1 in participants with ERBB2-mutated NSCLC with Brain Metastases (BM) and in participants with ERBB2-mutated or HER2-positive breast cancer with BM ± leptomeningeal disease (LMD)

SECONDARY OUTCOMES:
Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) [Part B and C] | Approximately 7 months
  Incidence and grade of Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs leading to dose modification in participants with ERBB2-mutated NSCLC with Brain Metastases (BM) and in participants with ERBB2-mutated or HER2-positive breast cancer with BM ± leptomeningeal disease (LMD)
Pharmacokinetics [Part A] | Approximately 28 days
  Area under the concentration-time curve (AUC) in participants with ERBB2 altered advanced solid tumors
Pharmacokinetics [Part A] | Approximately 28 days
  Maximum observed concentration (Cmax) in participants with ERBB2 altered advanced solid tumors
Pharmacokinetics [Part A] | Approximately 28 days
  Observed concentration at pre-dose (Ctrough)
Pharmacokinetics [Part A) | Approximately 28 days
  Time to measure concentration (Tmax)
Disease Response [Part A] | Approximately 6 months
  Overall objective response rate (ORR), as determined by confirmed complete response (CR) + confirmed partial response (PR) of all lesions (intracranial and extracranial) based on Investigator assessment using whole-body Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Disease Response [Part A] | Approximately 6 months
  Disease control rate (DCR), as determined by overall confirmed CR + confirmed PR + stable disease (SD) based on Investigator assessment using whole-body RECIST v1.1
Disease Response [Part B and Part C] | Approximately 6 months
  Disease Control Rate (DCR), determined by overall confirmed CR + confirmed PR +SD based on Investigator assessment using whole body RECIST v1.1
Disease Response [Part B and Part C] | Approximately 6 months
  Duration of Response (DOR), defined as time from first confirmed response (CR or PR) to the date of progressive disease (PD) or death from any cause, whichever occurs earlier
Disease Response [Part B and Part C] | Approximately 6 months
  Progression- free survival (PFS), defined as the time from the date of the first dose of study drug (Part B run-in and Part C)/ randomization (Part B randomized cohort) until the date of PD, based on Investigator assessment using whole body RECIST v1.1, or death from any cause, whichever comes earlier

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NEXT Oncology Texas, Austin, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia